CLINICAL TRIAL: NCT01376310
Title: MEK114375: A Rollover Study to Provide Continued Treatment With GSK1120212 to Subjects With Solid Tumors or Leukemia
Brief Title: GSK1120212 Rollover Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114375
Record Dates: First submitted 2011-02-03; First posted 2011-06-20 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — trametinib; Docetaxel; Erlotinib Hydrochloride; Pemetrexed; Carboplatin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Subjects on GSK1120212 Monotherapy who have been treated less than 24 weeks in their parent study.
  Interventions: Drug: GSK1120212
- Cohort B (Experimental): Subjects on GSK monotherapy who have been treated for 24 weeks or greater in their parent study. Also, subjects entering this study from any GSK1120212 combo trial.
  Interventions: Drug: GSK1120212; Drug: Docetaxel + GSK1120212; Drug: Erlotinib + GSK1120212; Drug: Pemetrexed + GSK1120212; Drug: Carboplatin + GSK1120212; Drug: Nab-paclitaxel + GSK1120212; Drug: Gemcitabine + GSK1120212; Drug: Everolimus + GSK1120212

INTERVENTIONS:
Drug: GSK1120212 — up to 2 mg/day
Drug: Docetaxel + GSK1120212 — dose as defined in the dose escalation protocol.
  Other Names: Taxotere
  Arms: Cohort B
Drug: Erlotinib + GSK1120212 — dose as defined in the dose escalation protocol.
  Other Names: Tarceva
  Arms: Cohort B
Drug: Pemetrexed + GSK1120212 — dose as defined in the dose escalation protocol
  Other Names: Alimta
  Arms: Cohort B
Drug: Carboplatin + GSK1120212 — dose as defined in the dose escalation protocol
  Other Names: Paraplatin
  Arms: Cohort B
Drug: Nab-paclitaxel + GSK1120212 — dose as defined in the dose escalation protocol
  Other Names: Abraxane
  Arms: Cohort B
Drug: Gemcitabine + GSK1120212 — dose as defined in the dose escalation protocol
  Other Names: Gemzar
  Arms: Cohort B
Drug: Everolimus + GSK1120212 — dose as defined in the dose escalation protocol
  Other Names: Afinitor
  Arms: Cohort B

SUMMARY:
This was an open-label study to permit subjects with solid tumors or leukemia, who were clinically benefitting on another GSK sponsored trial with GSK1120212 either monotherapy or in combination continued access to GSK1120212.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided signed informed consent for this study.
2. Has demonstrated compliance during the parent study with study treatment(s), treatment visit schedules, and the requirements and restrictions listed in the consent form.
3. Is currently participating in GSK1120212 study and is receiving treatment with GSK1120212.
4. Is currently receiving clinical benefit as determined by the investigator from previous treatment with GSK1120212 either as monotherapy or as part of a combination treatment regimen.
5. Continued ability to swallow and retain orally administered study treatment(s) and does not have any clinically significant GI abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
6. Female subjects of childbearing potential, as defined in the parent study, must be willing to continue practicing the same acceptable method of contraception as used in the parent study during the rollover study and for at least 4 months after the last dose of GSK1120212.
7. Female subjects of childbearing potential, as defined in parent study, must have negative serum pregnancy tests at the time of transition to this study.
8. Subjects enrolled in France: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

1. Permanent discontinuation of GSK1120212 in the parent study due to toxicity or disease progression.
2. Current use of a prohibitive medication(s) as listed in Section 6.2. NOTE: Use of anticoagulants such as warfarin is permitted; however, the international normalization ratio (INR) must be monitored in accordance with local institutional practice.
3. Any unresolved toxicity that meets the study treatment discontinuation or study withdrawal criteria from the parent study at the time of transition to this study.
4. Bazett-corrected QT (QTcB) interval ≥501 msec at the time of transition to this study
5. Left ventricular ejection fraction (LVEF) < institutional lower limit of normal (LLN) by ECHO (preferred) or MUGA scan at the time of transition to this study.
6. Nursing female.
7. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions at the time of transition to this study that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator or GSK Medical Monitor.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (13):
  - Novartis Investigative Site, Goodyear, Arizona
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, New Haven, Connecticut
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Tacoma, Washington
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Groningen, Netherlands
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 159 subjects received treatment with GSK1120212 and were included in the safety set.
Pre-assignment Details: Continued treatment with GSK1120212 was provided for subjects who had previously participated in a GSK1120212 study and who continued to receive clinical benefit as well as have an acceptable safety profile with GSK1120212.
Groups:
- Cohort A (GSK1120212 < 24 Weeks): Subjects on GSK1120212 Monotherapy and have been treated less than 24 weeks in their parent study.
- Cohort B (GSK1120212 >= 24 Weeks): Subjects on GSK monotherapy who have been treated for 24 weeks or greater in their parent study. Also, subjects entering this study from any GSK1120212 combo trial.
Period: Overall Study
Arm/Group | Cohort A (GSK1120212 < 24 Weeks) | Cohort B (GSK1120212 >= 24 Weeks)
Started | 126 | 33
Completed | 90 | 22
Not Completed | 36 | 11
Not completed — Study closed/terminated | 1 | 2
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Physician Decision | 26 | 7
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A (GSK1120212 < 24 Weeks) | Cohort B (GSK1120212 >= 24 Weeks) | Total
Number analyzed (Participants) | 126 | 33 | 159
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (12.34) | 61.7 (11.30) | 61.2 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 17 | 83
  Male | 60 | 16 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 116 | 28 | 144
  Black | 6 | 3 | 9
  Asian | 2 | 2 | 4
  Native American/Pacific Islander | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events as a measure of safety and tolerability
Time Frame: Until 30 days after the last dose of study treatment. Subjects may have continued to receive study treatment until disease progression, death, unacceptable toxicity or until locally commercially available. The maximum duration of exposure was 76 months.
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A (GSK1120212 < 24 Weeks) | Cohort B (GSK1120212 >= 24 Weeks)
Number analyzed (Participants) | 126 | 33
Participants
  Adverse Events | 119 | 30
  Treatment-Related Adverse Events | 101 | 26
  Serious Adverse Events | 26 | 13
  Treatment-Related Serious Adverse Events | 8 | 4

ADVERSE EVENTS:
Time Frame: From date of transition into this Rollover study until 30 days following the last dose (up to 76 months from date of transition).
Arm/Group | Cohort A (GSK1120212 < 24 Weeks) | Cohort B (GSK1120212 >= 24 Weeks)
All-Cause Mortality (participants affected / at risk) | 13/126 | 3/33
Serious Adverse Events (participants affected / at risk) | 26/126 | 13/33
Other Adverse Events (participants affected / at risk) | 115/126 | 28/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (GSK1120212 < 24 Weeks) (N=126) | Cohort B (GSK1120212 >= 24 Weeks) (N=33)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 1
Retinal vein occlusion (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 0 | 1
Moraxella infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Pyelonephritis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (GSK1120212 < 24 Weeks) (N=126) | Cohort B (GSK1120212 >= 24 Weeks) (N=33)
Anaemia (Blood and lymphatic system disorders) | 15 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 5
Ascites (Gastrointestinal disorders) | 5 | 2
Constipation (Gastrointestinal disorders) | 14 | 7
Diarrhoea (Gastrointestinal disorders) | 36 | 12
Dry mouth (Gastrointestinal disorders) | 13 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 33 | 7
Stomatitis (Gastrointestinal disorders) | 10 | 2
Vomiting (Gastrointestinal disorders) | 28 | 6
Chills (General disorders) | 10 | 2
Fatigue (General disorders) | 43 | 3
Mucosal inflammation (General disorders) | 7 | 4
Non-cardiac chest pain (General disorders) | 4 | 2
Oedema (General disorders) | 5 | 2
Oedema peripheral (General disorders) | 27 | 6
Pyrexia (General disorders) | 10 | 3
Cellulitis (Infections and infestations) | 3 | 2
Conjunctivitis (Infections and infestations) | 3 | 2
Folliculitis (Infections and infestations) | 0 | 2
Furuncle (Infections and infestations) | 0 | 2
Nail infection (Infections and infestations) | 2 | 2
Oral herpes (Infections and infestations) | 1 | 2
Paronychia (Infections and infestations) | 2 | 5
Pharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 6 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 2
Alanine aminotransferase increased (Investigations) | 8 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 1
Blood alkaline phosphatase increased (Investigations) | 7 | 1
Blood creatinine increased (Investigations) | 2 | 2
Weight decreased (Investigations) | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 18 | 2
Dehydration (Metabolism and nutrition disorders) | 14 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 2
Dizziness (Nervous system disorders) | 12 | 3
Dysgeusia (Nervous system disorders) | 8 | 1
Headache (Nervous system disorders) | 9 | 3
Migraine (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 35 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 4
Rash (Skin and subcutaneous tissue disorders) | 28 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 23 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 5 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2014-02-27): https://cdn.clinicaltrials.gov/large-docs/10/NCT01376310/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT01376310/SAP_001.pdf